CLINICAL TRIAL: NCT00979368
Title: Randomized, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BMS-816336 in Healthy Male Subjects
Brief Title: Safety Study of BMS-816336 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: MB124-001
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — BMS-816336

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- BMS-816336 or placebo (Panel 1) (Active Comparator)
  Interventions: Drug: BMS-816336; Drug: Placebo
- BMS-816336 or placebo (Panel 2) (Active Comparator)
  Interventions: Drug: BMS-816336; Drug: Placebo
- BMS-816336 or placebo (Panel 3) (Active Comparator)
  Interventions: Drug: BMS-816336; Drug: Placebo
- BMS-816336 or placebo (Panel 4) (Active Comparator)
  Interventions: Drug: BMS-816336; Drug: Placebo
- BMS-816336 or placebo (Panel 5) (Active Comparator)
  Interventions: Drug: BMS-816336; Drug: Placebo

INTERVENTIONS:
Drug: BMS-816336 — Suspension, Oral, 15 mg Active, Once on Day 1 only, 4 days
  Arms: BMS-816336 or placebo (Panel 1)
Drug: BMS-816336 — Suspension, Oral, 60 mg Active, Once on Day 1 only, 4 days
  Arms: BMS-816336 or placebo (Panel 2)
Drug: BMS-816336 — Suspension, Oral, 180 mg Active, Once on Day 1 only, 4 days
  Arms: BMS-816336 or placebo (Panel 3)
Drug: BMS-816336 — Suspension, Oral, 450 mg Active, Once on Day 1 only, 4 days
  Arms: BMS-816336 or placebo (Panel 4)
Drug: BMS-816336 — Suspension, Oral, 900 mg Active, Once on Day 1 only, 4 days
  Arms: BMS-816336 or placebo (Panel 5)
Drug: Placebo — Suspension, Oral, 0 mg, Once on Day 1 only, 4 days

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics following single oral doses of BMS-816336 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* BMI of 18 to 32 kg/m²
* Men only, ages 18-55 years

Exclusion Criteria:

* Sexually active men not using effective birth control if their partners are WOCBP
* Any significant acute or chronic medical illness
* Family history of Gilbert's disease
* History of Pancreatitis
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, EGG or clinical laboratory determinations
* QTc interval > 450 msec (corrected for heart rate using Fridericia's correction method, QTcF)
* Second- or third-degree A-V block or clinically relevant ECG abnormalities
* History of allergy to 11-β-HSD-1 inhibitors or related compounds
* Prior exposure to BMS-816336
* Use of St. John's Wort (Hypericum) within 4 weeks prior to the first dose of study drug and throughout the study
* Use of an oral, injectable, inhalable or suspension of glucocorticoid agents within 12 weeks of study drug administration
* Use of any glucocorticoid topical creams within 4 weeks of study drug administration
* Use of oral, injectable, or topical androgen agent within 12 weeks prior to enrollment

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Exposure to the investigational drug will be measured to assess safety and tolerability | Within 72 hours following dosing

SECONDARY OUTCOMES:
To assess the single dose Pharmacokinetics of BMS-816336 | During 72 hours following dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Melbourne, Victoria, Australia

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx